CLINICAL TRIAL: NCT02185339
Title: Effects of Deep Versus Moderate Neuromuscular Blockade on Intraoperative Respiratory Mechanics in Patients Undergoing Laparoscopic Renal Surgery: a Prospective, Randomized, Parallel Design Study
Brief Title: Effects of Deep Neuromuscular Blockade on Intraoperative Respiratory Mechanics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sanghyun Hong, Assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: dNMBonResp
Record Dates: First submitted 2014-06-27; First posted 2014-07-09 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Laparoscopic Renal Surgery; Laparoscopy; Muscle Relaxation
Keywords: Respiratory mechanics; Respiratory function test; Hemodynamics
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dNMB group (Experimental): For patients randomized to the dNMB group, intravenous infusion of 0.6 mg/kg/h rocuronium will be administered 10 minutes after the administration of intubation dose or after the return of post-tetanic count (PTC), whichever comes first. Then, the infusion rate will be titrated according to PTC (target to keep PTC between 1 to 2). Infusion rate will be increased or be reduced at a rate of 0.1 mg/kg/h if PTC is > or < than 1-2 to maintain deep muscle relaxation throughout the surgery. Neuromuscular monitoring will be carried out by monitoring the adductor pollicis muscle in response to ulnar nerve stimulation. A dose of sugammadex (4 mg/kg) will be administered at the end of the surgery. Patients will be extubated when the train of four ratio is ≥0.9.
  Interventions: Drug: Rocuronium
- mNMB group (Active Comparator): For patients randomized to the mNMB group, intravenous infusion of 0.2 mg/kg/h rocuronium will be administered 30 minutes after the administration of intubation dose or after the appearance of train-of-four (TOF) count >2, whichever comes first. Then, the infusion rate will be titrated according to TOF (target to keep TOF between 1 to 2). Infusion rate will be increased or reduced at a rate of 0.1 mg/kg/h if TOF is > or < than 1-2. A dose of sugammadex (2 mg/kg) will be administered at the end of the surgery. Patients will be extubated when the train of four ratio is ≥0.9.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Intravenous infusion rate of rocuronium will be titrated to keep post-tetanic count between 1 to 2.
  Other Names: Esmeron®
  Arms: dNMB group
Drug: Rocuronium — Intravenous infusion rate of rocuronium will be titrated to keep train-of-four count between 1 to 2.
  Other Names: Esmeron®
  Arms: mNMB group

SUMMARY:
The primary objective of the current study is to compare intraoperative respiratory mechanics in patients receiving laparoscopic renal surgery under deep neuromuscular blockade (dNMB) and under moderate neuromuscular blockade (mNMB). In addition, we will compare intraoperative hemodynamics and postoperative pulmonary function between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients scheduled to undergo laparoscopic renal surgery

Exclusion Criteria:

* BMI ≥35 kg/m2
* Known neuromuscular disease
* History of chronic obstructive pulmonary disease
* Asthma
* Pneumothorax
* Bronchopleural fistula
* Previous lung surgery
* Previous retroperitoneal surgery
* Hemodynamic instability
* History of cardiopulmonary disease
* Renal insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyun Hong, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at Seoul St. Mary's Hospital from July 2014 to January 2015.
Groups:
- Deep Neuromuscular Blockade (Deep NMB) Group: For patients randomized to the dNMB group, intravenous infusion of 0.6 mg/kg/h rocuronium was administered 10 minutes after the administration of intubation dose or after the return of post-tetanic count (PTC), whichever came first. Then, the infusion rate was titrated according to PTC (target to keep PTC between 1 and 2). Infusion rate was increased or be reduced at a rate of 0.1 mg/kg/h if PTC is > or < than 1-2 to maintain deep muscle relaxation throughout the surgery. Neuromuscular monitoring was carried out by monitoring the adductor pollicis muscle in response to ulnar nerve stimulation. A dose of sugammadex (4 mg/kg) was administered at the end of the surgery. Patients were extubated when the train of four ratio was ≥0.9.
- Moderate Neuromuscular Blockade (Moderate NMB) Group: For patients randomized to the mNMB group, intravenous infusion of 0.2 mg/kg/h rocuronium was administered 30 minutes after the administration of intubation dose or after the appearance of train-of-four (TOF) count, whichever came first. Then, the infusion rate was titrated according to TOF (target to keep TOF between 1 to 2). Infusion rate was increased or reduced at a rate of 0.1 mg/kg/h if TOF is > or < than 1-2. A dose of sugammadex (2 mg/kg) was administered at the end of the surgery. Patients were extubated when the train of four ratio was ≥0.9.
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (10.7) | 49.8 (11.0) | 49.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Thoracopulmonary Compliance
Description: Was measured with a patient spirometry monitor through a flow sensor.
  Measurements were obtained at the following four time points: (1) 15 min after a patient positioning in lateral decubitus before inducing the pneumoperitoneum (T Lateral); (2) 1 h after pneumoperitoneum induction with the patient in the lateral decubitus position (T Lat+PP1h); (3) 2 h after pneumoperitoneum induction with the patient in the lateral decubitus position (T Lat+PP2h); and (4) at the end of surgery, 15 min after abdominal deflation in the lateral decubitus position (T EndPP).
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: ml/cmH2O
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
ml/cmH2O
  T Lateral | 51.9 (9.8) | 52.3 (11.2)
  T Lat+PP1h | 34.6 (6.8) | 31.9 (6.2)
  T Lat+PP2h | 33.6 (7.7) | 30.8 (6.7)
  T EndPP | 54.1 (11.5) | 52.6 (11.7)

2. Secondary Outcome: Arterial Oxygen Tension/Inspired Oxygen Fraction
Description: Was calculated from arterial blood oxygen analysis. Measurements were obtained at (1) T Lateral, (2) T Lat+PP1h, (3) T Lat+PP2h, and (4) EndPP.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
mmHg
  T Lateral | 477 (100) | 483 (117)
  T Lat+PP1h | 467 (103) | 461 (90)
  T Lat+PP2h | 468 (86) | 465 (89)
  T EndPP | 493 (82) | 487 (79)

3. Secondary Outcome: Arterial to End-tidal Partial Pressure of Carbon Dioxide Difference
Description: Was calculated from arterial blood and expired carbon dioxide analysis. Measurements were obtained at (1) T Lateral, (2) T Lat+PP1h, (3) T Lat+PP2h, and (4) EndPP.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
mmHg
  T Lateral | 4.3 (1.7) | 4.3 (1.4)
  T Lat+PP1h | 5.8 (2.1) | 7.1 (2.2)
  T Lat+PP2h | 5.8 (2.6) | 7.2 (2.0)
  T EndPP | 4.2 (2.1) | 5.3 (2.4)

4. Secondary Outcome: Estimated Dead Space
Description: as for outcome 3
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: % of respiratory dead space
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
% of respiratory dead space
  T Lateral | 11.8 (4.6) | 11.9 (4.0)
  T Lat+PP1h | 14.1 (5.1) | 16.5 (4.7)
  T Lat+PP2h | 14.1 (6.1) | 16.4 (4.0)
  T EndPP | 12.0 (5.5) | 14.8 (6.2)

5. Secondary Outcome: Pulmonary Shunt
Description: Was calculated using the formula: pulmonary shunt = (pulmonary capillary oxygen content - arterial oxygen content) / (pulmonary capillary oxygen content - venous oxygen content). Pulmonary capillary oxygen partial pressure is assumed to be equal to alveolar oxygen partial pressure.
  Measurements were obtained at (1) T Lateral, (2) T Lat+PP1h, (3) T Lat+PP2h, and (4) EndPP.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: % of shunt
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
% of shunt
  T Lateral | 13.2 (5.2) | 12.4 (5.7)
  T Lat+PP1h | 12.7 (4.8) | 13.2 (6.2)
  T Lat+PP2h | 15.0 (8.9) | 14.8 (7.0)
  T EndPP | 11.9 (4.9) | 14.1 (6.7)

6. Other Pre Specified Outcome: Stroke Volume Variation
Description: Was calculated by taking '(maximum stroke volume - minimum stroke volume) / mean stroke volume' over a respiratory cycle using the FloTrac™ sensor and the Vigileo™ monitor.
  Measurements were obtained at (1) T Lateral, (2) T Lat+PP1h, (3) T Lat+PP2h, and (4) EndPP.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: % of mean stroke volume
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
% of mean stroke volume
  T Lateral | 9.2 (2.0) | 9.3 (1.4)
  T Lat+PP1h | 11.3 (3.3) | 12.9 (3.4)
  T Lat+PP2h | 11.4 (3.5) | 12.0 (2.6)
  T EndPP | 7.3 (2.5) | 7.9 (2.6)

7. Other Pre Specified Outcome: Cardiac Index
Description: Was obtained from arterial pressure waveform analysis using the FloTrac™ sensor and the Vigileo™ monitor.
  Measurements were obtained at (1) T Lateral, (2) T Lat+PP1h, (3) T Lat+PP2h, and (4) EndPP.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
L/min/m^2
  T Lateral | 2.4 (0.4) | 2.4 (0.5)
  T Lat+PP1h | 2.8 (1.0) | 2.6 (0.6)
  T Lat+PP2h | 2.9 (0.7) | 2.8 (0.6)
  T EndPP | 3.0 (0.8) | 3.1 (0.7)

8. Other Pre Specified Outcome: Surgical Condition
Description: Subjective rating of the view on the operating field was assessed by the surgeon who performed the surgery (optimal condition, good, acceptable, poor, extremely poor)
Time Frame: At completion of pneumoperitoneum surgery
Measure: Number; unit: Participants
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
Participants
  Extremely poor | 0 | 0
  Poor | 0 | 1
  Acceptable | 0 | 1
  Good | 1 | 7
  Optimal | 29 | 21

9. Other Pre Specified Outcome: Postoperative Pain
Description: Postoperative pain was measured by Visual Analogue Scale (VAS). Participants were asked to report their level of pain by pointing to a horizontal line, 10 cm in length. The scale (0-10 scores) was anchored by "no pain" (score of 0) and "pain as bad as it could be" (score of 10).
  Measurements were made at postoperative (PO) 1h, PO 2h, PO 6h, PO 24h, and PO 48h.
Time Frame: Postoperative 2 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Number analyzed (Participants) | 30 | 30
Scores on a scale
  PO 1h | 5.4 (2.0) | 5.9 (1.6)
  PO 2h | 5.1 (2.1) | 4.9 (1.6)
  PO 6h | 4.3 (2.3) | 4.5 (1.8)
  PO 24h | 2.2 (1.7) | 2.4 (1.8)
  PO 48h | 2.2 (1.7) | 2.4 (1.8)

ADVERSE EVENTS:
Arm/Group | Deep Neuromuscular Blockade (Deep NMB) Group | Moderate Neuromuscular Blockade (Moderate NMB) Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes